CLINICAL TRIAL: NCT00018564
Title: Novel Therapies for Essential Tremor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NEUD-048-00S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Therapeutics

INTERVENTIONS:
Drug: treatments for essential tremor

SUMMARY:
This clinical research program is designed to evaluate medications as new treatments for essential tremor. Essential tremor is a common condition with few available therapies.

DETAILED DESCRIPTION:
Each medication will be evaluated for effectiveness against tremor in a randomized, placebo-controlled, cross-over, double blind clinical research trial. Tremor will be assessed with accepted rating scales and accelerometry

ELIGIBILITY:
1. Diagnosis of essential tremor.
2. Tremor rating scale score 3 or one or both upper extremities
3. Unsatisfactory response to primidone or to propanolol
4. Not taking tremor-inducing drug
5. Able to comply with visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Fredricka Martin, Ph.D.
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States